CLINICAL TRIAL: NCT02394795
Title: A Phase III, Randomized, Controlled Study of mFOLFOX6 + Bevacizumab Combination Therapy Versus mFOLFOX6 + Panitumumab Combination Therapy in Chemotherapy-naive Patients With KRAS/NRAS Wild-type, Incurable/Unresectable, Advanced/Recurrent Colorectal Cancer
Brief Title: Panitumumab and RAS, Diagnostically-useful Gene Mutation for mCRC
Acronym: PARADIGM
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Takeda (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Panitumumab-3001; U1111-1164-9167 (Other: WHO); JapicCTI-142731 (Registry Identifier: JapicCTI); jRCTs031180246 (Registry Identifier: Japan Registry of Clinical Trials); UMIN000016776 (Registry Identifier: UMIN Clinical Trials Registry)
Record Dates: First submitted 2015-03-16; First posted 2015-03-20 (Estimated); Results first posted 2023-11-01 (Actual); Last update posted 2023-11-01 (Actual); Status verified 2023-01

CONDITIONS: Colorectal Cancer
Keywords: Metastatic colorectal cancer, Panitumumab, mFOLFOX6, Bevacizumab
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Oxaliplatin; Fluorouracil; Panitumumab; Bevacizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group P; mFOLFOX6 + panitumumab combination therapy (Experimental): OXA: 85 mg/m2/day 1 l-LV: 200 mg/m2/day 1 5-FU iv: 400 mg/m2/day 1 5-FU civ: 2400 mg/m2/day 1-3 panitumumab: 6 mg/kg mFOLFOX6 + panitumumab combination therapy, once every two weeks.
  Interventions: Drug: oxaliplatin (OXA), levofolinate calcium (l-LV), 5-FU, panitumumab
- Group B; mFOLFOX6 + bevacizumab combination therapy (Active Comparator): OXA: 85 mg/m2/day 1 l-LV: 200 mg/m2/day 1 5-FU iv: 400 mg/m2/day 1 5-FU civ: 2400 mg/m2/day 1-3 bevacizumab: 5 mg/kg/ mFOLFOX6 + bevacizumab combination therapy, once every two weeks.
  Interventions: Drug: oxaliplatin (OXA), levofolinate calcium (l-LV), 5-FU, bevacizumab

INTERVENTIONS:
Drug: oxaliplatin (OXA), levofolinate calcium (l-LV), 5-FU, panitumumab — oxaliplatin (OXA), levofolinate calcium (l-LV), panitumumab: intra-venous infusion 5-FU: bolus and continuous intra-venous infusion
  Arms: Group P; mFOLFOX6 + panitumumab combination therapy
Drug: oxaliplatin (OXA), levofolinate calcium (l-LV), 5-FU, bevacizumab — oxaliplatin (OXA), levofolinate calcium (l-LV), bevacizumab: intra-venous infusion 5-FU: bolus and continuous intra-venous infusion
  Arms: Group B; mFOLFOX6 + bevacizumab combination therapy

SUMMARY:
The purpose of this study is to verify the efficacy of mFOLFOX6 + panitumumab combination therapy and mFOLFOX6 + bevacizumab combination therapy in first-line treatment of chemotherapy-naive patients with KRAS/NRAS wild-type, incurable/unresectable, advanced/recurrent colorectal cancer.

DETAILED DESCRIPTION:
The purpose of this study is to verify the efficacy of mFOLFOX6 + panitumumab combination therapy and mFOLFOX6 + bevacizumab combination therapy in first-line treatment of chemotherapy-naive patients with KRAS/NRAS wild-type, incurable/unresectable, advanced/recurrent colorectal cancer.

This study will enroll a total of approximately 800 participants (400 per group).

Participants will be randomized to either the mFOLFOX6 + panitumumab arm (Group P) or mFOLFOX6 + bevacizumab arm (Group B) at 1:1 ratio at the time of registration.

Group P and Group B treatment regimen shown below should be administered once every two weeks, following dose, schedule and route of administration.

Group P; mFOLFOX6 + panitumumab combination therapy, once every two weeks OXA: 85 mg/m2/day 1 l-LV: 200 mg/m2/day 1 5-FU iv: 400 mg/m2/day 1 5-FU civ: 2400 mg/m2/day 1-3 panitumumab: 6 mg/kg

Group B; mFOLFOX6 + bevacizumab combination therapy, once every two weeks OXA: 85 mg/m2/day 1 l-LV: 200 mg/m2/day 1 5-FU iv: 400 mg/m2/day 1 5-FU civ: 2400 mg/m2/day 1-3 bevacizumab: 5 mg/kg

This trial is conducted by multicenter and is scheduled for 12 months as whole administration period.

ELIGIBILITY:
Inclusion Criteria:

1. Investigator and subinvestigator judge a candidate is understand clinical trial and comply this protocol.

   Investigator is those who participate in conducting a study and oversight the study duties at a site.
2. Patients who have given written consent to take part in the study after detailed explanation of the study prior to enrollment
3. Aged ≥20 to <80 years at the time of informed consent
4. Patients with unresectable adenocarcinoma originating in the large intestine (excluding carcinoma of the appendix and anal canal cancer)
5. Patients with lesion(s) that can be evaluated. It is not essential to be evaluated the tumor according to the RECIST ver. 1.1.
6. Patients who have not received chemotherapy for colorectal cancer. Patients who experience relapse more than 24 weeks (168 days) after the final dose of perioperative adjuvant chemotherapy with fluoropyrimidine agents may be enrolled. Patients who have received perioperative adjuvant chemotherapy including oxaliplatin are excluded.
7. Patients classified as KRAS/NRAS wild-type by KRAS/NRAS testing. KRAS/NRAS test will be performed using the in vitro diagnostic listed in the National Health Insurance.

   Patients with no mutation in any of the codons shown below are considered wild type. It is not considered wild type if either of the codons are not evaluable or not tested.

   KRAS: EXON2 (codon 12, 13), EXON3 (codon 59, 61), EXON4 (codon 117, 146) NRAS：EXON2 (codon 12, 13), EXON3 (codon 59, 61), EXON4 (codon 117, 146)
8. Patients who satisfy the following criteria for the major organ function in tests performed within 14 days prior to enrollment

   * Neutrophil count ≥ 1.5×10^3/µL
   * Platelet count ≥ 1.0×10^4/µL
   * Hemoglobin ≥ 9.0 g/dL
   * Total bilirubin ≤ 2.0 mg/dL
   * AST ≤ 100 IU/L (≤ 200 IU/L if liver metastases are present)
   * ALT ≤ 100 IU/L (≤ 200 IU/L if liver metastases are present)
   * Serum creatinine ≤ 1.5 mg/dL
   * PT-INR < 1.5 (< 3.0 for patients treated with oral warfarin)
   * Satisfies at least one of these conditions

     1. Urine protein (dip stick method) ≤ 1+
     2. UPC (urine protein creatinine) ratio ≤ 1.0
     3. Urinary protein ≤ 1000 mg/ 24hours
9. ECOG performance status (PS) of 0 or 1
10. Life expectancy of ≥ 3 months (90 days) after enrollment

Exclusion Criteria:

1. Radiotherapy received within 4 weeks (28 days) prior to enrollment. Treatments aimed at relieving pain for bone metastases are excluded.
2. Known brain metastasis or strongly suspected of brain metastasis
3. Synchronous cancers or metachronous cancers with a disease-free period of ≤ 5 years (excluding colorectal cancer) excluding mucosal cancers cured or be possibly cured by regional resection (esophageal, stomach, and cervical cancer, non-melanoma skin cancer, bladder cancer, etc.).
4. Body cavity fluid that requires treatment (pleural effusion, ascites, pericardial effusion, etc.)
5. Patients who do not want to use contraception to prevent pregnancy, and women who are pregnant or breast-feeding, or test positive for pregnancy
6. Nonhealing surgical wound (excluding implanted venous reservoirs)
7. Active hemorrhage requiring blood transfusion
8. Disease requiring systemic steroids for treatment (excluding topical steroids)
9. The patient who has placed colonic stent
10. Intestinal resection within 4 weeks prior to enrollment or colostomy within 2 weeks prior to enrollmentt
11. History or obvious and extensive CT findings of interstitial pulmonary disease (interstitial pneumonia, pulmonary fibrosis, etc.)
12. Patients with unstable angina, myocardial infarction, cerebral hemorrhage, arterial thromboembolism such as cerebral infarction, or have history of these desease less than 24 weeks (168 days) before registration (except for lacunar infarction asymptomatic)
13. Serious drug hypersensitivity
14. Local or systemic active infection requiring treatment, or fever indicating infection
15. NYHA class II or higher heart failure or serious heart disease
16. Intestinal paralysis, gastrointestinal obstruction, or uncontrollable diarrhoea (incapacitating symptoms despite adequate treatment)
17. Poorly controlled hypertension
18. Poorly controlled diabetes mellitus
19. Active hepatitis B
20. Known HIV infection
21. Peripheral neuropathy of ≥ Grade 2 by CTCAE (Japanese edition JCOG version 4.03)
22. Other patients judged by the investigator or subinvestigator to be ineligible for enrollment in the study (e.g. Patients who might agree to participate under compulsion).

Ages: 20 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 823 (Actual)
Dates: Start 2015-05-29 (Actual); Primary Completion 2022-01-14 (Actual); Study Completion 2022-01-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Takeda
Locations (154):
- Japan (154):
  - Ichinomiya, Aichi-ken
  - Komaki, Aichi-ken
  - Kōnan, Aichi-ken
  - Nagakute, Aichi-ken
  - Nagoya, Aichi-ken
  - Okazaki, Aichi-ken
  - Toyoake, Aichi-ken
  - Toyohashi, Aichi-ken
  - Toyokawa, Aichi-ken
  - Toyota, Aichi-ken
  - Yatomi, Aichi-ken
  - Daisen, Akita
  - Hirosaki, Aomori
  - Misawa, Aomori
  - Kashiwa, Chiba
  - Yachiyo, Chiba
  - Matsuyama, Ehime
  - Tōon, Ehime
  - Tsuruga, Fukui
  - Yoshida, Fukui
  - Kitakyushu, Fukuoka
  - Koga, Fukuoka
  - Kurume, Fukuoka
  - Omuta, Fukuoka
  - Aizu-Wakamatsu, Fukushima
  - Iwaki, Fukushima
  - Kōriyama, Fukushima
  - Shirakawa, Fukushima
  - Hashima, Gifu
  - Kakamigahara, Gifu
  - Minokamo, Gifu
  - Okazai, Gifu
  - Ōgaki, Gifu
  - Maebashi, Gunma
  - Ōta, Gunma
  - Fukuyama, Hiroshima
  - Hakodate, Hokkaido
  - Kitami, Hokkaido
  - Kushiro, Hokkaido
  - Obihiro, Hokkaido
  - Otaru, Hokkaido
  - Sapporo, Hokkaido
  - Akashi, Hyōgo
  - Amagasaki, Hyōgo
  - Himeji, Hyōgo
  - Kobe, Hyōgo
  - Nishinomiya, Hyōgo
  - Hitachi, Ibaraki
  - Kasama, Ibaraki
  - Ryūgasaki, Ibaraki
  - Tsuchiura, Ibaraki
  - Tsukuba, Ibaraki
  - Hakusan, Ishikawa-ken
  - Kaga, Ishikawa-ken
  - Kahoku, Ishikawa-ken
  - Kanazawa, Ishikawa-ken
  - Nanao, Ishikawa-ken
  - Morioka, Iwate
  - Kida, Kagawa-ken
  - Marugame, Kagawa-ken
  - Takamatsu, Kagawa-ken
  - Fujisawa, Kanagawa
  - Hiratsuka, Kanagawa
  - Isehara, Kanagawa
  - Kamakura, Kanagawa
  - Kanazawachō, Kanagawa
  - Sagamihara, Kanagawa
  - Yokohama, Kanagawa
  - Yokosuka, Kanagawa
  - Nankoku, Kochi
  - Matsuzaka, Mie-ken
  - Tsu, Mie-ken
  - Yokkaichi, Mie-ken
  - Ishinomaki, Miyagi
  - Murata, Miyagi
  - Natori-shi, Miyagi
  - Ōsaki, Miyagi
  - Sendai, Miyagi
  - Matsumoto, Nagano
  - Saku, Nagano
  - Ōmura, Nagasaki
  - Sasebo, Nagasaki
  - Ikoma, Nara
  - Tenri, Nara
  - Yamatotakada, Nara
  - Yufu, Oita Prefecture
  - Kurashiki, Okayama-ken
  - Naha, Okinawa
  - Tomigusuku, Okinawa
  - Urasoe, Okinawa
  - Hirakata, Osaka
  - Kawachi-Nagano, Osaka
  - Moriguchi, Osaka
  - Neyagawa, Osaka
  - Sayama, Osaka
  - Suita, Osaka
  - Kawagoe, Saitama
  - Kitaadachi, Saitama
  - Koshigaya, Saitama
  - Moriyama, Shiga
  - Ōtsu, Shiga
  - Izumi, Shimane
  - Izumo, Shimane
  - Hamamatsu, Shizuoka
  - Izunokuni, Shizuoka
  - Sunto, Shizuoka
  - Shimotsuga, Tochigi
  - Shimotsuke, Tochigi
  - Utsunomiya, Tochigi
  - Komatsushimachō, Tokushima
  - Bunkyo-ku, Tokyo
  - Chiyoda-ku, Tokyo
  - Chuo-ku, Tokyo
  - Itabashi-ku, Tokyo
  - Koto-ku, Tokyo
  - Machida, Tokyo
  - Meguro-ku, Tokyo
  - Minato-ku, Tokyo
  - Musashino, Tokyo
  - Ōta-ku, Tokyo
  - Shinagawa-ku, Tokyo
  - Shinjuku-ku, Tokyo
  - Yonago, Tottori
  - Kurobe-shi, Toyama
  - Takaoka, Toyama
  - Sakata, Yamagata
  - Tsuruoka, Yamagata
  - Iwakuni, Yamaguchi
  - Ube, Yamaguchi
  - Kofu, Yamanashi
  - Akita
  - Aomori
  - Chiba
  - Fukui
  - Fukuoka
  - Gifu
  - Ibaraki
  - Kagoshima
  - Kochi
  - Kumamoto
  - Kyoto
  - Miyazaki
  - Nagano
  - Nagasaki
  - Niigata
  - Okayama
  - Okinawa
  - Osaka
  - Saga
  - Saitama
  - Shizuoka
  - Tokushima
  - Toyama
  - Yamagata

IPD SHARING:
Plan to Share IPD: Yes
Takeda provides access to the de-identified individual participant data (IPD) for eligible studies to aid qualified researchers in addressing legitimate scientific objectives (Takeda's data sharing commitment is available on https://clinicaltrials.takeda.com/takedas-commitment?commitment=5). These IPDs will be provided in a secure research environment following approval of a data sharing request, and under the terms of a data sharing agreement.
Supporting Information: Study Protocol, SAP, ICF, CSR
Access Criteria: IPD from eligible studies will be shared with qualified researchers according to the criteria and process described on https://vivli.org/ourmember/takeda/. For approved requests, the researchers will be provided access to anonymized data (to respect patient privacy in line with applicable laws and regulations) and with information necessary to address the research objectives under the terms of a data sharing agreement.
URL: https://vivli.org/ourmember/takeda/

REFERENCES:
- [Derived] Shitara K, Muro K, Watanabe J, Yamazaki K, Ohori H, Shiozawa M, Takashima A, Yokota M, Makiyama A, Akazawa N, Ojima H, Yuasa Y, Miwa K, Yasui H, Oki E, Sato T, Naitoh T, Komatsu Y, Kato T, Mori I, Yamanaka K, Hihara M, Soeda J, Misumi T, Yamamoto K, Yamashita R, Akagi K, Ochiai A, Uetake H, Tsuchihara K, Yoshino T. Baseline ctDNA gene alterations as a biomarker of survival after panitumumab and chemotherapy in metastatic colorectal cancer. Nat Med. 2024 Mar;30(3):730-739. doi: 10.1038/s41591-023-02791-w. Epub 2024 Feb 12. PMID 38347302
- [Derived] Watanabe J, Muro K, Shitara K, Yamazaki K, Shiozawa M, Ohori H, Takashima A, Yokota M, Makiyama A, Akazawa N, Ojima H, Yuasa Y, Miwa K, Yasui H, Oki E, Sato T, Naitoh T, Komatsu Y, Kato T, Hihara M, Soeda J, Misumi T, Yamamoto K, Akagi K, Ochiai A, Uetake H, Tsuchihara K, Yoshino T. Panitumumab vs Bevacizumab Added to Standard First-line Chemotherapy and Overall Survival Among Patients With RAS Wild-type, Left-Sided Metastatic Colorectal Cancer: A Randomized Clinical Trial. JAMA. 2023 Apr 18;329(15):1271-1282. doi: 10.1001/jama.2023.4428. PMID 37071094
- [Derived] Yoshino T, Uetake H, Tsuchihara K, Shitara K, Yamazaki K, Oki E, Sato T, Naitoh T, Komatsu Y, Kato T, Yamanaka K, Iwasaki K, Soeda J, Hihara M, Yamanaka T, Ochiai A, Muro K. Rationale for and Design of the PARADIGM Study: Randomized Phase III Study of mFOLFOX6 Plus Bevacizumab or Panitumumab in Chemotherapy-naive Patients With RAS (KRAS/NRAS) Wild-type, Metastatic Colorectal Cancer. Clin Colorectal Cancer. 2017 Jun;16(2):158-163. doi: 10.1016/j.clcc.2017.01.001. Epub 2017 Jan 24. PMID 28237539
- See also: To obtain more information on the study, click here/on this link — https://clinicaltrials.takeda.com/study-detail/5f6b60294db2bf003ab499d1

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in the study at 197 investigative sites in Japan from 29 May 2015 to 14 January 2022.
Pre-assignment Details: Participants with KRAS/NRAS wild-type, incurable/unresectable, advanced/recurrent colorectal cancer were enrolled and randomized to either the mFOLFOX6 + panitumumab arm (Group P) or mFOLFOX6 + bevacizumab arm (Group B) at 1:1 ratio.
Period: Overall Study
Arm/Group | Group P; mFOLFOX6 + Panitumumab Combination Therapy | Group B; mFOLFOX6 + Bevacizumab Combination Therapy
Started | 404 | 407
Completed | 1 | 1
Not Completed | 403 | 406
Not completed — Adverse Event | 92 | 70
Not completed — Lost to Follow-up | 0 | 1
Not completed — Withdrawal by Subject | 17 | 26
Not completed — Lack of Efficacy | 181 | 211
Not completed — Death | 4 | 5
Not completed — Physician Decision | 109 | 93

BASELINE CHARACTERISTICS:
Population: Full analysis set (FAS): all randomized patients who received at least one dose of protocol treatment without major protocol deviation.
Groups:
- Total: Total of all reporting groups
Arm/Group | Group P; mFOLFOX6 + Panitumumab Combination Therapy | Group B; mFOLFOX6 + Bevacizumab Combination Therapy | Total
Number analyzed (Participants) | 400 | 402 | 802
Age, Customized [Count of Participants; unit: Participants]
  65 years old or over | 236 | 234 | 470
  64 years old or less | 164 | 168 | 332
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 148 | 134 | 282
  Male | 252 | 268 | 520
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 400 | 402 | 802
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  Japan | 400 | 402 | 802
Number of Participants with Primary Tumor Categorized by Location [Count of Participants; unit: Participants] — Reported data were number of participants with primary tumor location categorized by Left side, Right side, or the Other at the start of this study. Primary tumor site (left side/right side/other) defined as following. Left side: Single lesion or multiple lesions in the descending colon, sigmoid colon, rectosigmoid region, or rectum. Right side: Single lesion or multiple lesions in the cecum, ascending colon, or transverse colon. Other: Multiple primary tumors extending over the right and left sides.
  Participants
    Left side | 312 | 292 | 604
    Right side | 84 | 103 | 187
    Other | 4 | 7 | 11
Medical History [Count of Participants; unit: Participants] — Medical history defined as a disease or a health condition for each participant before start of the study. Medical history was classified as congenital anomalies, hematologic disorders, psychiatric and nervous system disorders, cardiovascular disorders, respiratory disorders, GI disorders, hepatic and biliary disorders, renal disease and other medical history. Other medical history included all medical history except for those mentioned above.
  Participants
    Had No Medical History | 86 | 78 | 164
    Had Medical History | 314 | 324 | 638
Medical Complications [Count of Participants; unit: Participants] — Complications defined as a disease or a health condition for each participant at the start of study. Complications were classified as congenital anomalies, endocrine disorders, hematologic disorders, psychiatric and nervous system disorders, cardiovascular disorders, respiratory disorders, gastrointestinal (GI) disorders, renal disease and other complications.
  Participants
    Had No Medical Complications | 162 | 159 | 321
    Had Medical Complications | 238 | 243 | 481
Eastern Cooperative Oncology Group (ECOG) Performance Status (PS) [Count of Participants; unit: Participants] — ECOG assessed participant's performance status on 5 point scale: 0=Fully active/able to carry on all pre-disease activities without restriction; 1=restricted in physically strenuous activity but ambulatory/able to carry out light or sedentary work; 2=ambulatory (>50 percent of waking hours), capable of all self-care but unable to carry out any work activities; 3=capable of only limited self-care, confined to bed/chair >50 percent of waking hours; 4=completely disabled, cannot carry on any self-care, totally confined to bed/chair.
  Participants
    0 | 328 | 319 | 647
    1 | 71 | 83 | 154
    2 | 1 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: OS in Participants With Left-sided Tumors
Description: OS was measured as the time from the date of randomization to the date of death due to any cause. The left-sided tumors were defined as primary tumors occupying a left-sided site include the descending colon, sigmoid colon, and rectum.
Time Frame: Up to approximately 60 months
Population: Full analysis set (FAS): all randomized patients who received at least one dose of protocol treatment without major protocol deviation. The number analyzed is the number of participants with data available for analysis.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Group P; mFOLFOX6 + Panitumumab Combination Therapy | Group B; mFOLFOX6 + Bevacizumab Combination Therapy
Number analyzed (Participants) | 312 | 292
Months | 37.85 [34.10 to 42.58] | 34.30 [30.92 to 40.28]

2. Primary Outcome: Overall Survival (OS) in All Participants
Description: OS was measured as the time from the date of randomization to the date of death due to any cause.
Time Frame: Up to approximately 60 months
Population: as for baseline characteristics
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Group P; mFOLFOX6 + Panitumumab Combination Therapy | Group B; mFOLFOX6 + Bevacizumab Combination Therapy
Number analyzed (Participants) | 400 | 402
Months | 36.24 [32.03 to 39.03] | 31.28 [29.27 to 34.10]

3. Secondary Outcome: Progression-Free Survival (PFS) in Participants With Left-sided Tumors
Description: PFS was defined as the time from the date of randomization to the earlier of Progressive Disease (PD) per Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1 or death due to any cause. The left-sided tumors were defined as primary tumors occupying a left-sided site include the descending colon, sigmoid colon, and rectum.
Time Frame: Up to approximately 60 months
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Group P; mFOLFOX6 + Panitumumab Combination Therapy | Group B; mFOLFOX6 + Bevacizumab Combination Therapy
Number analyzed (Participants) | 312 | 292
Months | 13.70 [12.65 to 15.34] | 13.24 [11.40 to 14.49]

4. Secondary Outcome: Progression-Free Survival (PFS) in All Participants
Description: PFS was defined as the time from the date of randomization to the earlier of Progressive Disease (PD) per Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1 or death due to any cause.
Time Frame: Up to approximately 60 months
Population: as for baseline characteristics
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Group P; mFOLFOX6 + Panitumumab Combination Therapy | Group B; mFOLFOX6 + Bevacizumab Combination Therapy
Number analyzed (Participants) | 400 | 402
Months | 12.91 [11.30 to 13.63] | 11.99 [11.30 to 13.47]

5. Secondary Outcome: Response Rate (RR) in All Participants
Description: RR was defined as number of participants who achieve Complete Response (CR) and Partial Response (PR) as the best overall response per RECIST version 1.1.The best overall response was CR, followed by PR, stable disease (SD), progressive disease (PD), and not evaluable (NE). CR: disappearance of all target lesions. Any pathological lymph nodes must have reduction in short axis to <10 mm. PR: at least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum diameters as the best overall response after randomization., SD: neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD, taking as reference the smallest sum diameters while on study. PD: at least a 20% increase in the sum of diameters of target lesions, taking as reference the smallest sum on study (this includes the baseline sum if that is the smallest on study).
Time Frame: Up to approximately 60 months
Population: Full analysis set (FAS): all randomized patients who received at least one dose of protocol treatment without major protocol deviation. The number analyzed is the number of participants with data available for analysis. RR was assessed in participants with evaluable lesions at baseline.
Measure: Count of Participants; unit: Participants
Arm/Group | Group P; mFOLFOX6 + Panitumumab Combination Therapy | Group B; mFOLFOX6 + Bevacizumab Combination Therapy
Number analyzed (Participants) | 394 | 397
Participants
  CR | 11 | 14
  PR | 284 | 253
  SD | 79 | 112
  PD | 20 | 18

6. Secondary Outcome: Duration of Response (DOR)
Description: DOR means that the period from the day when either CR or PR is first confirmed until the day of documented PD or the day of death due to all causes, whichever occurs earlier.
Time Frame: Up to approximately 60 months
Population: Full analysis set (FAS): all randomized patients who received at least one dose of protocol treatment without major protocol deviation. The number analyzed is the number of participants with data available for analysis. DOR was evaluated in participants with complete or partial response.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Group P; mFOLFOX6 + Panitumumab Combination Therapy | Group B; mFOLFOX6 + Bevacizumab Combination Therapy
Number analyzed (Participants) | 295 | 267
Months | 11.86 [10.51 to 13.37] | 10.74 [9.46 to 12.19]

7. Secondary Outcome: Number of Participants Treated With Curative Surgical Resection After Chemotherapy
Description: Curative surgical resection was defined as complete resection.
Time Frame: Up to approximately 60 months
Population: Full analysis set (FAS): all randomized patients who received at least one dose of protocol treatment without measure protocol deviation.
Measure: Count of Participants; unit: Participants
Arm/Group | Group P; mFOLFOX6 + Panitumumab Combination Therapy | Group B; mFOLFOX6 + Bevacizumab Combination Therapy
Number analyzed (Participants) | 400 | 402
Participants | 66 | 44

8. Secondary Outcome: Number of Participants With Treatment-emergent Adverse Events (TEAE)
Description: Adverse event (AE) was defined as any untoward medical occurrence in a participant administered a pharmaceutical product and which did not necessarily have a causal relationship with this treatment. A TEAE was defined as an adverse event with an onset that occurred in the treatment period after receiving the protocol treatment.
Time Frame: Up to approximately 60 months
Population: Safety analysis set (SAS): all patients who initiated the protocol treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Group P; mFOLFOX6 + Panitumumab Combination Therapy | Group B; mFOLFOX6 + Bevacizumab Combination Therapy
Number analyzed (Participants) | 404 | 407
Participants | 402 | 398

ADVERSE EVENTS:
Time Frame: Up to approximately 60 months
Description: At each visit the investigator had to document any occurrence of adverse events and abnormal laboratory findings. Any event spontaneously reported by the participant or observed by the investigator was recorded, irrespective of the relation to study treatment.
Arm/Group | Group P; mFOLFOX6 + Panitumumab Combination Therapy | Group B; mFOLFOX6 + Bevacizumab Combination Therapy
All-Cause Mortality (participants affected / at risk) | 14/404 | 9/407
Serious Adverse Events (participants affected / at risk) | 115/404 | 95/407
Other Adverse Events (participants affected / at risk) | 399/404 | 392/407
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Group P; mFOLFOX6 + Panitumumab Combination Therapy (N=404) | Group B; mFOLFOX6 + Bevacizumab Combination Therapy (N=407)
Anaemia (Blood and lymphatic system disorders) | 2 | 1
Disseminated intravascular coagulation (Blood and lymphatic system disorders) | 0 | 1
Febrile neutropenia (Blood and lymphatic system disorders) | 3 | 1
Pancytopenia (Blood and lymphatic system disorders) | 1 | 0
Angina pectoris (Cardiac disorders) | 1 | 0
Atrial fibrillation (Cardiac disorders) | 1 | 1
Cardiac failure (Cardiac disorders) | 1 | 0
Hypothyroidism (Endocrine disorders) | 1 | 0
Cataract (Eye disorders) | 0 | 1
Rhegmatogenous retinal detachment (Eye disorders) | 1 | 0
Abdominal distension (Gastrointestinal disorders) | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 1 | 2
Anal haemorrhage (Gastrointestinal disorders) | 0 | 1
Ascites (Gastrointestinal disorders) | 0 | 1
Constipation (Gastrointestinal disorders) | 1 | 2
Diaphragmatic hernia (Gastrointestinal disorders) | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 5 | 2
Duodenal perforation (Gastrointestinal disorders) | 1 | 0
Enterocolitis (Gastrointestinal disorders) | 3 | 1
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 0
Gastrointestinal perforation (Gastrointestinal disorders) | 0 | 1
Haemorrhoidal haemorrhage (Gastrointestinal disorders) | 1 | 0
Haemorrhoids (Gastrointestinal disorders) | 1 | 0
Ileus (Gastrointestinal disorders) | 3 | 7
Inguinal hernia (Gastrointestinal disorders) | 1 | 0
Intestinal obstruction (Gastrointestinal disorders) | 3 | 3
Large intestinal obstruction (Gastrointestinal disorders) | 0 | 1
Large intestinal stenosis (Gastrointestinal disorders) | 0 | 1
Large intestine perforation (Gastrointestinal disorders) | 1 | 3
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 1
Mechanical ileus (Gastrointestinal disorders) | 3 | 2
Melaena (Gastrointestinal disorders) | 1 | 0
Nausea (Gastrointestinal disorders) | 3 | 3
Pneumatosis intestinalis (Gastrointestinal disorders) | 1 | 0
Small intestinal obstruction (Gastrointestinal disorders) | 0 | 1
Stomatitis (Gastrointestinal disorders) | 2 | 1
Vomiting (Gastrointestinal disorders) | 1 | 1
Death (General disorders) | 1 | 1 — The reasons of events are not determined because assessment findings were insufficient to specify the reason.
Fatigue (General disorders) | 1 | 0
Implant site dehiscence (General disorders) | 0 | 1
Malaise (General disorders) | 3 | 1
Mucosal inflammation (General disorders) | 0 | 1
Pyrexia (General disorders) | 3 | 3
Sudden death (General disorders) | 0 | 1 — The reasons of events are not determined because assessment findings were insufficient to specify the reason.
Bile duct stenosis (Hepatobiliary disorders) | 0 | 2
Bile duct stone (Hepatobiliary disorders) | 2 | 1
Cholangitis (Hepatobiliary disorders) | 4 | 2
Cholecystitis acute (Hepatobiliary disorders) | 0 | 1
Hepatic failure (Hepatobiliary disorders) | 0 | 2
Jaundice (Hepatobiliary disorders) | 1 | 0
Jaundice cholestatic (Hepatobiliary disorders) | 0 | 1
Primary biliary cholangitis (Hepatobiliary disorders) | 0 | 1
Anaphylactic reaction (Immune system disorders) | 3 | 2
Anaphylactic shock (Immune system disorders) | 1 | 0
Hypersensitivity (Immune system disorders) | 3 | 0
Abdominal abscess (Infections and infestations) | 2 | 0
Abdominal wall abscess (Infections and infestations) | 0 | 1
Anal abscess (Infections and infestations) | 0 | 1
Anorectal infection (Infections and infestations) | 0 | 1
Bacteraemia (Infections and infestations) | 0 | 1
Cellulitis (Infections and infestations) | 0 | 1
Device related infection (Infections and infestations) | 3 | 4
Diverticulitis (Infections and infestations) | 0 | 1
Enteritis infectious (Infections and infestations) | 1 | 1
Herpes zoster (Infections and infestations) | 1 | 0
Infection (Infections and infestations) | 1 | 0
Influenza (Infections and infestations) | 1 | 0
Liver abscess (Infections and infestations) | 1 | 0
Muscle abscess (Infections and infestations) | 1 | 0
Pelvic abscess (Infections and infestations) | 1 | 0
Peritonitis (Infections and infestations) | 3 | 1
Pneumonia (Infections and infestations) | 6 | 3
Pneumonia bacterial (Infections and infestations) | 1 | 2
Pneumonia pneumococcal (Infections and infestations) | 0 | 2
Pyelonephritis (Infections and infestations) | 1 | 1
Renal abscess (Infections and infestations) | 0 | 1
Sepsis (Infections and infestations) | 1 | 2
Subcutaneous abscess (Infections and infestations) | 0 | 1
Urinary tract infection (Infections and infestations) | 1 | 2
Vascular device infection (Infections and infestations) | 1 | 1
Ankle fracture (Injury, poisoning and procedural complications) | 0 | 1
Compression fracture (Injury, poisoning and procedural complications) | 1 | 0
Fracture (Injury, poisoning and procedural complications) | 1 | 0
Hip fracture (Injury, poisoning and procedural complications) | 1 | 1
Humerus fracture (Injury, poisoning and procedural complications) | 0 | 1
Infusion related reaction (Injury, poisoning and procedural complications) | 0 | 1
Pelvic fracture (Injury, poisoning and procedural complications) | 1 | 0
Pneumothorax traumatic (Injury, poisoning and procedural complications) | 0 | 1
Postoperative ileus (Injury, poisoning and procedural complications) | 0 | 1
Spinal compression fracture (Injury, poisoning and procedural complications) | 7 | 1
Spinal fracture (Injury, poisoning and procedural complications) | 0 | 1
Stoma complication (Injury, poisoning and procedural complications) | 0 | 1
Stoma site dermatitis (Injury, poisoning and procedural complications) | 1 | 0
Stoma site inflammation (Injury, poisoning and procedural complications) | 0 | 1
Urinary tract stoma complication (Injury, poisoning and procedural complications) | 0 | 1
Vascular access complication (Injury, poisoning and procedural complications) | 0 | 1
Wound complication (Injury, poisoning and procedural complications) | 0 | 1
C-reactive protein increased (Investigations) | 1 | 0
Neutrophil count decreased (Investigations) | 1 | 1
White blood cell count decreased (Investigations) | 1 | 0
White blood cell count increased (Investigations) | 1 | 0
Decreased appetite (Metabolism and nutrition disorders) | 14 | 9
Dehydration (Metabolism and nutrition disorders) | 4 | 0
Electrolyte imbalance (Metabolism and nutrition disorders) | 1 | 0
Hyperammonaemia (Metabolism and nutrition disorders) | 2 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 1 | 0
Hypernatraemia (Metabolism and nutrition disorders) | 1 | 0
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 | 1
Hypocalcaemia (Metabolism and nutrition disorders) | 1 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 1 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 2 | 0
Hypomagnesaemia (Metabolism and nutrition disorders) | 1 | 0
Malnutrition (Metabolism and nutrition disorders) | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 | 0
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 1 | 0
Osteoporosis (Musculoskeletal and connective tissue disorders) | 1 | 0
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 3
Metastases to central nervous system (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Rectal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Thyroid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Altered state of consciousness (Nervous system disorders) | 1 | 0
Cerebral haemorrhage (Nervous system disorders) | 1 | 0
Cerebral infarction (Nervous system disorders) | 1 | 0
Depressed level of consciousness (Nervous system disorders) | 2 | 0
Dizziness (Nervous system disorders) | 1 | 0
Encephalopathy (Nervous system disorders) | 0 | 1
Epilepsy (Nervous system disorders) | 1 | 0
Headache (Nervous system disorders) | 0 | 1
Hepatic encephalopathy (Nervous system disorders) | 0 | 1
Subarachnoid haemorrhage (Nervous system disorders) | 1 | 0
Anxiety (Psychiatric disorders) | 1 | 0
Acute kidney injury (Renal and urinary disorders) | 2 | 1
Hydronephrosis (Renal and urinary disorders) | 0 | 3
Ureterolithiasis (Renal and urinary disorders) | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 11 | 5
Lung disorder (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pulmonary artery thrombosis (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 3 | 3
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Tracheal stenosis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Upper respiratory tract inflammation (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 1 | 0
Drug eruption (Skin and subcutaneous tissue disorders) | 1 | 0
Skin disorder (Skin and subcutaneous tissue disorders) | 1 | 0
Aortic aneurysm (Vascular disorders) | 0 | 1
Deep vein thrombosis (Vascular disorders) | 3 | 2
Embolism (Vascular disorders) | 2 | 0
Jugular vein thrombosis (Vascular disorders) | 1 | 0
Venous thrombosis limb (Vascular disorders) | 0 | 2
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Group P; mFOLFOX6 + Panitumumab Combination Therapy (N=404) | Group B; mFOLFOX6 + Bevacizumab Combination Therapy (N=407)
Anaemia (Blood and lymphatic system disorders) | 37 | 50
Constipation (Gastrointestinal disorders) | 92 | 105
Diarrhoea (Gastrointestinal disorders) | 146 | 135
Nausea (Gastrointestinal disorders) | 158 | 160
Stomatitis (Gastrointestinal disorders) | 249 | 165
Vomiting (Gastrointestinal disorders) | 43 | 50
Fatigue (General disorders) | 158 | 162
Malaise (General disorders) | 63 | 66
Pyrexia (General disorders) | 25 | 48
Hypersensitivity (Immune system disorders) | 21 | 48
Nasopharyngitis (Infections and infestations) | 10 | 22
Paronychia (Infections and infestations) | 210 | 20
Alanine aminotransferase increased (Investigations) | 37 | 28
Aspartate aminotransferase increased (Investigations) | 38 | 32
Neutrophil count decreased (Investigations) | 201 | 224
Platelet count decreased (Investigations) | 86 | 80
White blood cell count decreased (Investigations) | 32 | 44
Decreased appetite (Metabolism and nutrition disorders) | 216 | 203
Hypokalaemia (Metabolism and nutrition disorders) | 31 | 8
Hypomagnesaemia (Metabolism and nutrition disorders) | 120 | 7
Neuropathy peripheral (Nervous system disorders) | 21 | 30
Peripheral sensory neuropathy (Nervous system disorders) | 286 | 300
Taste disorder (Nervous system disorders) | 125 | 94
Proteinuria (Renal and urinary disorders) | 9 | 31
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 2 | 21
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 13 | 80
Alopecia (Skin and subcutaneous tissue disorders) | 47 | 48
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 301 | 13
Dry skin (Skin and subcutaneous tissue disorders) | 186 | 38
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 94 | 57
Pruritus (Skin and subcutaneous tissue disorders) | 36 | 12
Rash (Skin and subcutaneous tissue disorders) | 41 | 15
Hypertension (Vascular disorders) | 7 | 76

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The first study related publication will be a multi-center publication submitted within 24 months after conclusion or termination of a study at all sites. After such multi site publication, all proposed site publications and presentations will be submitted to sponsor for review 60 days in advance of publication.

Site will remove Sponsor confidential information unrelated to study results. Sponsor can delay a proposed publication for another 60 days to preserve intellectual property.

DOCUMENTS (2):
  • Study Protocol (2022-01-05): https://cdn.clinicaltrials.gov/large-docs/95/NCT02394795/Prot_000.pdf
  • Statistical Analysis Plan (2022-02-03): https://cdn.clinicaltrials.gov/large-docs/95/NCT02394795/SAP_001.pdf